CLINICAL TRIAL: NCT04123522
Title: Using the High Resolution Impedance Manometry to Evaluate Swallowing Function After Cervical Spine Surgery: Anterior vs Posterior Approach
Brief Title: Using the High Resolution Impedance Manometry to Evaluate Swallowing Function After Cervical Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907079RINA
Record Dates: First submitted 2019-10-06; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Pharyngeal Pressure Change

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anterior cervical spine surgery: The patients will be enrolled for elective anterior cervical spine surgery.
  Interventions: Procedure: anterior approach
- posterior cervical spine surgery: The patients will be enrolled for elective postieor cervical spine surgery
  Interventions: Procedure: posterior appraoch

INTERVENTIONS:
Procedure: anterior approach — anterior approach
  Other Names: anterior appraoch
  Groups: anterior cervical spine surgery
Procedure: posterior appraoch — posteiror appraoch
  Other Names: posterior approach
  Groups: posterior cervical spine surgery

SUMMARY:
Dysphagia is a well-known complication following cervical spine surgery, including anterior or posterior approach. However, which muscle at oropharyngeal region weakness and the recovery course of these patients are still unknown.

The high resolution impedance manometry (HRIM) could be used to measure the postoperative recovery esophageal function.

DETAILED DESCRIPTION:
Dysphagia is a well-known complication following cervical spine surgery, including anterior or posterior approach. However, which muscle at oropharyngeal region weakness and the recovery course of these patients are still unknown.

The high resolution impedance manometry (HRIM) could be used to measure the postoperative recovery esophageal function.

In this study, using the high resolution impedance manometry to determine (1) whether the occurrence of dysphagia in the postoperative 1 or 7 days and 1 month in the patients receiving anterior vs posterior approach of cervical spine surgery (2) which muscle in the pharyngeal region would be destroyed Consecutive patients who will fulfill the criteria of cervical spine surgery patients under general anesthesia and aged >= 20 will be enrolled. The patients would receive the dysphagia questionnaire. All subjects would receive the swallowing function by HRIM before the surgeries. The cough test was also measured. After the surgery, the patient would be followed the swallowing function in the postoperative one day, and 1 week by HRIM and questionnaire.

This study would expect (1) that the posterior cervical spine surgery would result in dysphagia greater than baseline, but less than that of anterior cervical procedures; (2) decreasing upper esophageal sphincter (UES) pressure may be the reason of postoperative dysphagia in the anterior cervical spine surgery, resulted from the intraoperative traction; (3) decreasing hypopharyngeal muscle pressure may be the reason of postoperative dysphagia in the posterior spine surgery, resulted from the prone and flexion positioning.

ELIGIBILITY:
Inclusion Criteria:1. Patients who fulfill the criteria of cervical spine surgery under general anesthesia 2. Aged from 20-80 years old -

Exclusion Criteria:

- 1. Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.

2. Patients who have the risk of difficult ventilation or intubation. 3. pregnant women 4. coagulopathy

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients recieved elective cervical spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-11-02 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
mean pharyngeal peak pressure | preoperative, postoperative day 1 and 7
  the pharyngeal presssure change during swallowing

IPD SHARING:
Plan to Share IPD: No